CLINICAL TRIAL: NCT00931307
Title: Evaluation of Lotrafilcon A Lenses Over a Three Month Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-335-C-013
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2010-10-06 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2010-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

ARMS (1):
- Lotrafilcon A (Experimental)
  Interventions: Device: Lotrafilcon A contact lens

INTERVENTIONS:
Device: Lotrafilcon A contact lens — Silicone hydrogel, spherical, soft contact lens

SUMMARY:
The purpose of this trial is to assess the performance of a Lotrafilcon A contact lens over a 3-month period.

ELIGIBILITY:
Inclusion Criteria:

* On examination, have ocular findings considered to be "normal" and which would not prevent a subject from safely wearing contact lenses.
* Be willing and able to follow instructions and meet the schedule of follow-up visits as defined in the informed consent.
* Be able to wear the study lenses in the available powers.
* Currently wear contact lenses for a minimum of 5 days a week, and at least 8 hours a day.
* Other protocol inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment for this trial.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in an ophthalmic clinical trial.
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Any use of medications for which contact lens wear would be contraindicated, in the opinion of the investigator.
* History of corneal refractive surgery.
* Other protocol inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Lotrafilcon A: Silicone hydrogel, spherical, experimental soft contact lenses worn on the same basis as habitual contact lenses as prescribed by eye care practitioner
Period: Overall Study
Arm/Group | Lotrafilcon A
Started | 22
Completed | 9
Not Completed | 13
Not completed — Lack of Efficacy | 12
Not completed — Biomicroscopy | 1

BASELINE CHARACTERISTICS:
Groups:
- Lotrafilcon A: Silicone hydrogel, spherical, soft contact lens
Arm/Group | Lotrafilcon A
Number analyzed (Participants) | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 32.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Comfort After Insertion
Description: Comfort after insertion of contact lens (30 seconds to 1 minute), as interpreted by the subject and reported by the subject as a single, retrospective evaluation of 3-month's wear time. Comfort after insertion was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 3 months
Population: Per protocol. Analysis excluded major protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: Scale of 1 to 10
Arm/Group | Lotrafilcon A
Number analyzed (Participants) | 9
Scale of 1 to 10 | 7.9 (1.6)

ADVERSE EVENTS:
Time Frame: Duration of trial: 4 months
Arm/Group | Lotrafilcon A
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
Due to the small number of subjects successfully completing this trial, the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.